CLINICAL TRIAL: NCT05392101
Title: Low Dose Iron Chelation as TReatment of Oxidative Damage in Patients With Sickle Cell Disease: the TROS Study
Brief Title: Low Dose Iron Chelation as TReatment of Oxidative Damage in Sickle Cell Disease
Acronym: TROS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Erfan Nur, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021_007
Record Dates: First submitted 2022-01-25; First posted 2022-05-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Deferasirox

STUDY DESIGN:
Intervention Model Description: Phase II open label interventional pilot study. It is a mono-center cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient group: 360mg deferasirox (Experimental): Patient group receiving treatment
  Interventions: Drug: Deferasirox 360 MG

INTERVENTIONS:
Drug: Deferasirox 360 MG — Deferasirox 360 MG p.o. once daily
  Other Names: Exjade

SUMMARY:
Objective:

To study the safety and efficacy of deferasirox as treatment of oxidative stress in adult subjects with sickle cell disease.

Endpoints:

The investigators will determine whether treatment with iron chelators results in decreased sickling of RBCs, oxidative stress, neutrophil activation, inflammation, endothelial activation and hypercoagulability and ultimately reduced disease severity. If the hypothesis is confirmed in this pilot dose-finding study, a larger randomized controlled clinical trial will be initiated.

Study design:

This will be an open-label pilot study, including 12 patients per dose group with a maximum of 3 dose groups. As the antioxidant capacity of deferasirox might be dose-dependent, the investigators will start with the highest dose of deferasirox (360 mg) deemed adequate for chronic use without causing iron depletion in adult SCD patients.

Study population:

Adult patients with sickle cell anemia (HbSS) or HbS-β0-thalassemia (HbSβ0-thal) visiting the outpatient-clinic of the Academic Medical Center, Amsterdam will be asked for inclusion in the study.

DETAILED DESCRIPTION:
Rationale:

Sickle cell disease (SCD) is an inherited hemoglobinopathy, characterized by hemolysis, vaso-occlusive crises and organ damage resulting in reduced life expectancy. Oxidative stress is a major pathophysiological factor in SCD playing a significant role in the SCDrelated microvascular dysfunction, vaso-occlusion, inflammation and organ damage. Chronic life-long intravascular hemolysis with the resulting excessive levels of cell-free heme and iron is the major cause of increased production of reactive oxygen species (ROS) in SCD. The cell-free heme rapidly releases its iron which is the main driving force of redox reactions. The hydrophobic heme also rapidly intercalates into the plasma membrane of (endothelial) cells where it releases its iron. This potentiates cell damage by catalyzing non-enzymatic generation of ROS. By inactivating NO, cell-free ferrous hemoglobin reduces nitric oxide (NO) bioavailability, limiting the important vasodilative, anti-thrombotic and anti-inflammatory properties of NO. Since the ongoing and unremitting release of iron is the major cause of oxidative stress in SCD, it is imminent to investigate the role of iron chelators as antioxidative therapy in this disease. Iron chelators have been shown to protect various cells, including red blood cells (RBCs) and endothelial cells, against oxidative toxicity. The investigators recently found that sequestration of free iron by the iron-chelator deferoxamine blocked activation of neutrophils and their release of neutrophil extracellular traps (NETs) by sera of SCD patients (preliminary data). NETs have been demonstrated to be toxic, especially, to endothelial cells. In this study the investigators will test the hypothesis that treating sickle cell patients with low doses of readily available iron chelators might reduce oxidative stress by capturing the excessively released intravascular cell-free iron.

Objective:

To study the safety and efficacy of deferasirox as treatment of oxidative stress in adult subjects with sickle cell disease.

Study design:

This will be an open-label pilot study, including 12 patients per dose group with a maximum of 3 dose groups. As the antioxidant capacity of deferasirox might be dose-dependent, the investigators will start with the highest dose of deferasirox (360 mg) deemed adequate for chronic use without causing iron depletion in adult SCD patients. Depending on the results, the investigators will continue with a following 6 weeks of treatment with a reduced dose (180mg once daily). One of the criteria for continuation of the study with a dose reduction is that least 3 of the 12 patients have to show a decrease of at least 25% in PoS or one of the main secondary endpoints. Another criterion is confirmation of the before seen good safety profile. Patients with results are offered to continue with the lower dose after a washout period of at least 4 weeks, this is not obliged. After this potential second dose phase of 180mg, the same process of result evaluation will take place to determine potential benefits of continuing with a second dose reduction of 90 mg deferasirox once daily. Again including the interested responding patients (after a washout period of at least 4 weeks). The study will be closed if <3 patients show a response in at least one of the endpoints. Also, if ≥ 4 patients in a dose group show iron depletion the study team will stop inclusion and treatment for that dose and continue to the next (lower) dose, excluding the depleted patients and continuing with patients that had no side effects after a washout of 4 weeks.

Study population:

Adult patients with sickle cell anemia (HbSS) or HbS-β0-thalassemia (HbSβ0-thal) visiting the outpatient-clinic of the Academic Medical Center, Amsterdam will be asked for inclusion in the study.

Intervention:

Once daily deferasirox, starting with the highest dose of 360 mg per day during 6 weeks. If positive results on study endpoints are observed (in at least 25% of participants) and low adverse events rates are seen the dose can be reduced to 180 mg (for 6 weeks) and potentially to 90mg (for 6 weeks).

Main study parameters/endpoints:

The main endpoints of this study are safety and efficacy. The investigators will evaluate safety by analysis of adverse events, medication use and physical and laboratory examinations.The primary efficacy endpoint will be the effect of deferasirox on sickling of red blood cells, measured as changes in Point of Sickling (PoS), as quantified by Oxygenscan. Other efficacy endpoints include the proportion of patients with decreases in hemoglobin S (HbS) %, oxidative stress as reflected by advanced glycation end-products (AGEs), decreased neutrophil activation, decreased endothelial activation and decreased in vitro adhesion of red blood cells and neutrophils.

Sample size analysis The primary aim of this pilot study is to obtain preliminary estimates of the mean and standard deviation of Point of Sickling (PoS). Data from (at least) 12 patients will enable us to estimate the mean and standard deviation of changes in PoS as a result of treatment with deferasirox and obtain a two-sided, 95% confidence interval for the mean change that will extend 0.566 times the standard deviation on both sides of the estimated mean change.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The risks of participation in this study are predicted to be very low. Deferasirox is a drug that has been widely used for years with good safety profile. The doses usually used are much higher 720 - 1430 mg daily than the intended doses in this study (360 - 90 mg). The investigators therefore do not expect to encounter the previously described side effects such as diarrhoea, decreased renal function, which are mostly dose-dependent. Patients will have to take study medication once a day for a period of 6 weeks. Patients will visit the outpatient clinic at baseline (T0) and then after 2 (T1), 4 (T2) and 6 (T3) weeks during the treatment. At 10 weeks (4 weeks after cessation of the study drug) patients will be seen for a final follow-up (T4). Blood samples will be drawn at all the above mentioned visits to monitor for therapeutic effects and potential side effects. Patients with positive effects of study medication, can be asked to participate in another cycle of 6 weeks in a lower dose.

ELIGIBILITY:
Inclusion criteria In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. High performance liquid chromatography confirmed diagnosis of HbSS or HbSβ0 genotype.
2. Aged 18-65 years
3. Written informed consent

Exclusion criteria A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Blood transfusion in the preceding four months
2. Already using iron chelation due to iron overload
3. Ferritin levels of <50 µg/L and/or transferrin saturation of < 0.20.
4. LDH of < 300 U/L
5. Pregnancy or the desire to get pregnant in the following 6 months
6. Impaired renal function of GFR < 60 ml/min/1,73m2(CKD-EPI), or chronic medication that influences renal function
7. Known allergic reaction to deferasirox.
8. Other somatic or cognitive condition disturbing adherence to study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Point of sickling | 4 months up to 8 months
  Point of sickling measures by oxygen scan. To measure deformability of Red Blood Cells in shear stress, during oxygen-depletion
Oxidative stress | 4 months up to 8 months
  Oxidative stress measured by AGES

CONTACTS AND LOCATIONS:
Overall Officials: Erfan Nur, MD, PHD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdan UMC location AMC, Amsterdam, Meibergdreef 9, Netherlands

IPD SHARING:
Plan to Share IPD: No